CLINICAL TRIAL: NCT05346263
Title: Efficacy of Intermittent Abdominal Pressure Ventilation in Neuromuscular Patients: Multicentre, Randomised Controlled Trial
Brief Title: Efficacy of Intermittent Abdominal Pressure Ventilation in Neuromuscular Patients
Acronym: IAPV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19/2021/CE_FdG/FC/SA
Record Dates: First submitted 2022-04-13; First posted 2022-04-26 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-03

CONDITIONS: Neuromuscular Diseases
Keywords: Neuromuscular Diseases;; Intermittent Abdominal Pressure Ventilation;; IAPV;
MeSH Terms: conditions — Neuromuscular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Abdominal Pressure Ventilation (Experimental): Patients in experimental group will be adapted to Intermittent Abdominal Pressure Ventilation (IAPV). Abdominal ventilation replaces part of usual ventilation (non invasive ventilation with mouthpiece or nasal-pillow)
  Interventions: Device: Intermittent Abdominal Pressure Ventilation
- Usual ventilation (Active Comparator): Patients in control group continue with usual ventilation (NIV through mouthpiece or nasal-pillow)
  Interventions: Device: Usual ventilation

INTERVENTIONS:
Device: Intermittent Abdominal Pressure Ventilation — Patients of experimental group will use IAPV in daytime ventilation. Intermittent abdominal pressure ventilation (IAPV) is a portable ventilator with an internal battery and PneumoBelt corset as an interface.
  Other Names: IAPV
  Arms: Intermittent Abdominal Pressure Ventilation
Device: Usual ventilation — NIV
  Arms: Usual ventilation

SUMMARY:
Non-Invasive Ventilation (NIV) is an established treatment to manage respiratory muscles dysfunction in neuromuscular disease, preventing the progression of respiratory failure to intubation and/or a tracheotomy. NIV is commonly needed at first during the night, but when the disease worsens, it is required during the day. It is provided via nasal or oronasal masks, causing discomfort and/or aesthetic issues that result in poor compliance.

Intermittent Abdominal Pressure Ventilation (IAPV) is a valid, though unconventional, alternative to daytime NIV: it consists of a portable ventilator with an internal battery and a corset as interface. The IAPV corset is lightweight, comfortable and, thanks to velcro fasteners, easier and better fitting than a face mask. Cyclical inflation of a rubber bladder inside the corset moves the diaphragm upwards like a pneumobelt causing air to enter in the lungs via the upper airways as gravity draws the diaphragm back to its resting position.

IAPV is indicated in neuromuscular disease and has already been tested in few preliminary studies and case reports. This study wants to verify the hypothesis of its application in population of neuromuscular patients.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Neuromuscular Disease (Amyotrophic Lateral Sclerosis, Duchenne Muscular Dystrophy, Spinal Muscular Atrophy, Pompe Disease)
* Non Invasive Ventilation > 16 hours/day
* Informed consent signed

Exclusion Criteria:

- Diagnosis of kyphoscoliosis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Blood Gas Analysis | 12 months
  Changes of respiratory parameters in terms of normalization of oxyemia (Arterial Pressure of oxygen 80-100 mmHg) and normalization of capnia (Arterial Pressure of carbon dioxide 35-45 mmHg), assessed by blood gas analysis

SECONDARY OUTCOMES:
Therapy adherence | 12 months
  Adherence to IAPV tested with Beliefs about Ventilation Questionnaire (BVQ). BVQ is a qualitative questionnaire: it consist of 25 items, where higher scores mean a better outcome.
Patients satisfaction to IAPV | 12 months
  Satisfaction to IAPV tested with Visual Analog Scale (VAS), with a score that ranges between 0 and 10, where a higher score means a worse outcome.
Caregivers satisfaction to IAPV | 12 months
  Satisfaction to IAPV tested with Visual Analog Scale (VAS), with a score that ranges between 0 and 10, where a higher score means a worse outcome.
Amelioration of Quality of life | 12 months
  Improvement of quality of life tested with World Health Organization Quality of Life-Brief (WHOQOL-Brief), with a score ranging from 0 to 100 for each of the four domain and where a higher score means a better outcome

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS S. Maria Nascente - Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No